CLINICAL TRIAL: NCT07029425
Title: Effectiveness of Manual Therapy in the Treatment of Attention Deficit Hyperactivity Disorder
Acronym: MT-ADHD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JJ JIMENEZ-REJANO (Other)
Responsible Party: Sponsor-Investigator, JJ JIMENEZ-REJANO, Director, University of Seville
Organization: University of Seville (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USeville-PFB
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Attention Deficit Hyperactivity Disorder; manual therapy; pediatrics
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: craniosacral therapy techniques. (Experimental): Experimental:
  Participants in the experimental group will receive Manual Therapy (MT) designed for this study, which will include craniosacral therapy techniques. The sessions will last 40 minutes and will be conducted twice a week for the first 4 weeks, followed by once a week for the final 4 weeks.
  Interventions: Procedure: Procedure: craniosacral therapy techniques.
- Control: placebo comparator. (Placebo Comparator): Sham Comparator:
  The placebo group will receive a dummy treatment with a duration of 40min, twice a week for the firt 4 week, follwed by once a week for the final 4 week.
  Interventions: Procedure: Placebo Group

INTERVENTIONS:
Procedure: Procedure: craniosacral therapy techniques. — Participants in the experimental group will receive Manual Therapy (MT) designed for this study, which will include craniosacral therapy techniques. The sessions will last 40 minutes and will be conducted twice a week for the first 4 weeks, followed by once a week for the final 4 weeks.
  Arms: Experimental: craniosacral therapy techniques.
Procedure: Placebo Group — The placebo group will receive a dummy treatment with a duration of 40min, twice a week for the firt 4 week, follwed by once a week for the final 4 week.
  Arms: Control: placebo comparator.

SUMMARY:
The main objective is to determine whether Manual Therapy (MT), in addition to conventional treatment, is more effective in improving ADHD symptoms than the application of conventional treatment alone.

DETAILED DESCRIPTION:
Background ADHD is a disorder that affects attention, behavior control, and emotions in children. Although medication and behavioral therapy can help, not all children respond well or may experience side effects, which leads to the search for alternative options. This disorder affects the daily lives of both the child and their family, and in adulthood, it can cause emotional, social, and work-related problems. Treatment usually includes medication, cognitive-behavioral therapy, parent training, and techniques such as mindfulness. A newer option is manual therapy (MT), which uses massage and craniosacral therapy to support the nervous system and improve emotional and behavioral regulation. Although some studies have shown promising results, more research is needed to confirm its effectiveness.

Materials and Methods: A randomized clinical trial will be conducted. The minimum sample size required for statistical significance is 60 subjects, divided into two groups with 30 participants each. The primary variable will be hyperactivity and attention deficit, assessed using the Conners Parent Rating Scale and the Conners Teacher Rating Scale. The secondary variable will be mood, measured using a facial expression scale.

Objetives To determine whether the addition of manual therapy to conventional treatment is more effective in improving ADHD symptoms than conventional treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed ADHD diagnosis according to DSM-5 criteria.
* Children and adolescents aged 6 to 12 years.
* Availability to attend all Manual Therapy (MT) sessions.
* Informed consent signed by legal guardians.

Exclusion Criteria:

* Severe concomitant psychiatric or neurological disorders (e.g., epilepsy, severe autism spectrum disorder, schizophrenia).
* Medical conditions that contraindicate MT (e.g., fractures, severe scoliosis, connective tissue diseases).
* Recent use of or changes in ADHD medication within the past 4 weeks.
* Simultaneous participation in other interventional studies.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Symptoms of ADHD (Parents Rating Scale) | At the star of the study (at basilne, 0 week), After the 2nd session (at the end of the first week), after 12th session (at the end of the eight week) and 4 months from the last session (24th week).
  Conners Parents Rating Scale. 48 items 0 = Never, 1 = Sometimes, 2 = Often, and 3 = Very Often. Scores 0-144. Scores greater than or equal to 59 = normal range, Scores 60-64 = mildly elevated symptom severity, Scores 65-69 = moderately elevated severity Scores > 70 = presence of highly elevated severity.
Symptoms of ADHD (Teacher Rating Scale) | At the star of the study (at basilne, 0 week), After the 2nd session (at the end of the first week), after 12th session (at the end of the eight week) and 4 months from the last session (24th week).
  Conners Teacher Rating Scale. 28 items. 0 = Never, 1 = Sometimes, 2 = Often, and 3 = Very Often. Scores 0-84. Scores greater than or equal to 59 = normal range, Scores 60-64 = mildly elevated symptom severity, Scores 65-69 = moderately elevated severity Scores > 70 = presence of highly elevated severity.

SECONDARY OUTCOMES:
Mood | At the star of the study (at basilne, 0 week), After the 2nd session (at the end of the first week), after 12th session (at the end of the eight week) and 4 months from the last session (24th week).
  Facial Expression Scale. It represents expressions from sadness (scored with 1) to happiness (scored with 4).

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo de Investigación Área de Fisioterapia CTS 305 - Universidad de Sevilla, Sevilla, Spain 41009, Alcalá de Henares, Madrid, Spain

REFERENCES:
- [Background] Chan SKC, Zhang D, Bogels SM, Chan CS, Lai KYC, Lo HHM, Yip BHK, Lau ENS, Gao TT, Wong SYS. Effects of a mindfulness-based intervention (MYmind) for children with ADHD and their parents: protocol for a randomised controlled trial. BMJ Open. 2018 Nov 12;8(11):e022514. doi: 10.1136/bmjopen-2018-022514. PMID 30420347
- [Background] Accorsi A, Lucci C, Di Mattia L, Granchelli C, Barlafante G, Fini F, Pizzolorusso G, Cerritelli F, Pincherle M. Effect of osteopathic manipulative therapy in the attentive performance of children with attention-deficit/hyperactivity disorder. J Am Osteopath Assoc. 2014 May;114(5):374-81. doi: 10.7556/jaoa.2014.074. PMID 24778002
- [Background] Danckaerts M, Sonuga-Barke EJ, Banaschewski T, Buitelaar J, Dopfner M, Hollis C, Santosh P, Rothenberger A, Sergeant J, Steinhausen HC, Taylor E, Zuddas A, Coghill D. The quality of life of children with attention deficit/hyperactivity disorder: a systematic review. Eur Child Adolesc Psychiatry. 2010 Feb;19(2):83-105. doi: 10.1007/s00787-009-0046-3. Epub 2009 Jul 26. PMID 19633992
- [Background] Crouzet L, Gramond A, Suehs C, Fabbro-Peray P, Abbar M, Lopez-Castroman J. Third-generation cognitive behavioral therapy versus treatment-as-usual for attention deficit and hyperactivity disorder: a multicenter randomized controlled trial. Trials. 2022 Jan 28;23(1):83. doi: 10.1186/s13063-021-05983-2. PMID 35090544
- [Background] Bellato A, Arora I, Hollis C, Groom MJ. Is autonomic nervous system function atypical in attention deficit hyperactivity disorder (ADHD)? A systematic review of the evidence. Neurosci Biobehav Rev. 2020 Jan;108:182-206. doi: 10.1016/j.neubiorev.2019.11.001. Epub 2019 Nov 10. PMID 31722229
- [Background] Polanczyk G, de Lima MS, Horta BL, Biederman J, Rohde LA. The worldwide prevalence of ADHD: a systematic review and metaregression analysis. Am J Psychiatry. 2007 Jun;164(6):942-8. doi: 10.1176/ajp.2007.164.6.942. PMID 17541055
- [Background] Robertz AC, Tornhage CJ, Nilsson S, Nyman V, Kantzer AK. Positive effects of tactile massage for adolescents with Attention Deficit/Hyperactivity Disorder (ADHD) - A small scale study. Complement Ther Clin Pract. 2024 Nov;57:101909. doi: 10.1016/j.ctcp.2024.101909. Epub 2024 Sep 25. PMID 39332064
- [Background] Musser ED, Backs RW, Schmitt CF, Ablow JC, Measelle JR, Nigg JT. Emotion regulation via the autonomic nervous system in children with attention-deficit/hyperactivity disorder (ADHD). J Abnorm Child Psychol. 2011 Aug;39(6):841-52. doi: 10.1007/s10802-011-9499-1. PMID 21394506
- [Background] Duric NS, Assmus J, Gundersen D, Duric Golos A, Elgen IB. Multimodal treatment in children and adolescents with attention-deficit/hyperactivity disorder: a 6-month follow-up. Nord J Psychiatry. 2017 Jul;71(5):386-394. doi: 10.1080/08039488.2017.1305446. Epub 2017 Mar 27. PMID 28345387
- [Background] Steinau S. Diagnostic Criteria in Attention Deficit Hyperactivity Disorder - Changes in DSM 5. Front Psychiatry. 2013 May 30;4:49. doi: 10.3389/fpsyt.2013.00049. eCollection 2013. No abstract available. PMID 23755024
- [Background] Pumprla J, Howorka K, Groves D, Chester M, Nolan J. Functional assessment of heart rate variability: physiological basis and practical applications. Int J Cardiol. 2002 Jul;84(1):1-14. doi: 10.1016/s0167-5273(02)00057-8. PMID 12104056
- [Background] Rechberger V, Biberschick M, Porthun J. Effectiveness of an osteopathic treatment on the autonomic nervous system: a systematic review of the literature. Eur J Med Res. 2019 Oct 25;24(1):36. doi: 10.1186/s40001-019-0394-5. PMID 31653268
- [Background] Mizuno Y, Cai W, Supekar K, Makita K, Takiguchi S, Tomoda A, Menon V. Methylphenidate remediates aberrant brain network dynamics in children with attention-deficit/hyperactivity disorder: A randomized controlled trial. Neuroimage. 2022 Aug 15;257:119332. doi: 10.1016/j.neuroimage.2022.119332. Epub 2022 May 28. PMID 35640787
- [Background] Haugan AJ, Sund AM, Young S, Thomsen PH, Lydersen S, Novik TS. Cognitive behavioural group therapy as addition to psychoeducation and pharmacological treatment for adolescents with ADHD symptoms and related impairments: a randomised controlled trial. BMC Psychiatry. 2022 Jun 2;22(1):375. doi: 10.1186/s12888-022-04019-6. PMID 35655149
- [Background] Cai W, Mizuno Y, Tomoda A, Menon V. Bayesian dynamical system analysis of the effects of methylphenidate in children with attention-deficit/hyperactivity disorder: a randomized trial. Neuropsychopharmacology. 2023 Oct;48(11):1690-1698. doi: 10.1038/s41386-023-01668-3. Epub 2023 Jul 25. PMID 37491674
- [Background] Cade A, Jones K, Holt K, Penkar AM, Haavik H. The Effects of Spinal Manipulation on Oculomotor Control in Children with Attention Deficit Hyperactivity Disorder: A Pilot and Feasibility Study. Brain Sci. 2021 Aug 6;11(8):1047. doi: 10.3390/brainsci11081047. PMID 34439666
- [Background] Bayo-Tallon V, Esquirol-Caussa J, Pamias-Massana M, Planells-Keller K, Palao-Vidal DJ. Effects of manual cranial therapy on heart rate variability in children without associated disorders: Translation to clinical practice. Complement Ther Clin Pract. 2019 Aug;36:125-141. doi: 10.1016/j.ctcp.2019.06.008. Epub 2019 Jul 2. PMID 31383430
- [Background] LeBaron S, Zeltzer L. Assessment of acute pain and anxiety in children and adolescents by self-reports, observer reports, and a behavior checklist. J Consult Clin Psychol. 1984 Oct;52(5):729-38. doi: 10.1037//0022-006x.52.5.729. No abstract available. PMID 6501658
- [Background] Pan MR, Dong M, Zhang SY, Liu L, Li HM, Wang YF, Qian QJ. One-year follow-up of the effectiveness and mediators of cognitive behavioural therapy among adults with attention-deficit/hyperactivity disorder: secondary outcomes of a randomised controlled trial. BMC Psychiatry. 2024 Mar 16;24(1):207. doi: 10.1186/s12888-024-05673-8. PMID 38491411
- [Background] Zhu C. Effects of Musicotherapy Combined with Cognitive Behavioral Intervention on the Cognitive Ability of Children with Attention Deficit Hyperactivity Disorder. Psychiatr Danub. 2022 Summer;34(2):288-295. doi: 10.24869/psyd.2022.288. PMID 35772139